CLINICAL TRIAL: NCT04563260
Title: Effect of Palonosetron on Effect-site Concentration of Remifentanil for Preventing Emergence Cough During General Anesthesia in Female Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Effect of Palonosetron on Remifentanil for Preventing Emergence Cough in Female
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Eun Kim, associate professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AJIRB-MED-THE-20-174
Record Dates: First submitted 2020-09-15; First posted 2020-09-24 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Gallbladder Diseases
MeSH Terms: conditions — Gallbladder Diseases | interventions — Saline Solution; Palonosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Control group receives the intravenous normal saline 2 mL.
  Interventions: Drug: Normal saline injection
- Palonosetron group (Experimental): Palonosetron group receives the intravenous palonosetron 1.5 mL (0.075 mg) + normal saline 0.5 mL.
  Interventions: Drug: Palonosetron Injection [Aloxi]

INTERVENTIONS:
Drug: Normal saline injection — Normal saline 2 mL, intravenous injection
  Arms: Control group
Drug: Palonosetron Injection [Aloxi] — Palonosetron 1.5 mL (0.075 mg) + Normal saline 0.5 mL, intravenous injection
  Arms: Palonosetron group

SUMMARY:
The primary purpose of this study is to investigate the optimal Ce of remifentanil for preventing emergence cough following extubation during general anesthesia in female patients who receive the palonosetron or not.

DETAILED DESCRIPTION:
Remifentanil is a potent ultrashort-acting opioid, with rapid onset and offset of drug effect. It allows rapid anesthetic emergence even after a prolonged infusion, and decreases the at-risk time during extubation. In addition, cough suppression of remifentanil enables smooth extubation with reduced complications. However, the infusion of remifentanil suppresses the emergence cough effectively in clinical practice, whereas it still delays the awakening from anesthesia, resulting in prolonged emergence time. Reduced Ce of remifentanil during emergence would decrease the adverse events that are associated with remifentanil infusion.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic cholecystectomy under general anesthesia

Exclusion Criteria:

* BMI > 30 kg/m2, respiratory infection, uncontrolled hypertension

Ages: 19 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
optimal Ce of remifentanil | From the end of surgery until the time of endotracheal extubation, about 20 minutes
  Using Dixon methods, evaluating of optimal Ce of remifentanil for preventing emergence cough following extubation during general anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine, Suwon, South Korea